CLINICAL TRIAL: NCT05418387
Title: A Pilot Social Network and Support Intervention to Improve Kidney and Liver Cancer Treatment Among Hispanics in Arizona
Brief Title: A Social Support Intervention to Improve Treatment Among Hispanic Kidney and Liver Cancer Patients in Arizona
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study will be withdrawn as the Principal Investigator, Ken Batai, left the institution prior to study activation.
Sponsor: University of Arizona (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 35185
Record Dates: First submitted 2022-06-01; First posted 2022-06-14 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Renal Cell Carcinoma; Hepatocellular Carcinoma
Keywords: Kidney cancer; Renal cell carcinoma; Hepatocellular carcinoma; Social support; Social network; Caregiver; Hispanics
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients randomized to receive the Social Support Network intervention
  Interventions: Behavioral: Social Support Network Intervention
- Patient Navigation (Active Comparator): Patients randomized to receive Usual Care (patient navigation)
  Interventions: Behavioral: Control (Patient Navigation Service)

INTERVENTIONS:
Behavioral: Social Support Network Intervention — The navigator will provide basic patient navigation services and Supportive Health Education to the patient/caregiver dyads in the patient's preferred language using the Support Network Workbook. The intervention will consist of 7 telephone sessions. There will be 2 sessions in the first month and one session per month after the first month (6 months total). Coaching and guiding techniques rather than lectures will be used applying dyads' specific social support network information. Each session will be about 30 minutes long.
  Arms: Group A
Behavioral: Control (Patient Navigation Service) — The patient navigator will provide basic patient navigation services consisting of health care barriers/social needs assessment, referral to social workers (if eligible) and support groups for patients and caregivers, and transportation assistance without Supportive Health Education. Patient/caregiver dyads in the control group will be contacted at 3- and 6-months post-enrollment and asked about their experience receiving treatment, any challenges they encountered or are currently facing, and the care support they received from family members, friends, CHWs, and health care providers.
  Arms: Patient Navigation

SUMMARY:
This project will develop and pilot test social support intervention for an underserved population, Hispanics in Arizona, who have high rates of kidney and liver cancer to improve health equity. The investigators will incorporate caregivers (family members) and other individuals in a patient's social network in survivorship, who are especially critical to quality cancer care. Caregivers provide more than half the care to cancer survivors and are often instrumental in facilitating the survivor to receive the care needed and adhere to guidelines. Through this project, the investigators will be able to leverage the resources of the Cancer Heath Equity Research Center (e.g., community outreach) to develop an intervention that has the potential for scalability and reach and recruit a sufficient sample across the target catchment area (including rural participants who may live near the US-Mexico border).

DETAILED DESCRIPTION:
The goals of this 6-month patient navigator implemented telephone-based social support intervention are to assess 1) feasibility of a full-scale intervention in Hispanic kidney and liver cancer patients and 2) the effect of intervention on timely treatment initiation and adherence to follow-up care in (n=100). The pilot intervention in this study will determine effective recruitment and study participant retention strategies, intervention feasibility and acceptability, and best timing to initiate the intervention, length of intervention, and required sample size.

The primary outcome of this pilot intervention is to assess feasibility of a full-scale intervention study by determining: 1) how many patients are screened and enrolled per month, 2) how many enrolled patients participate in each intervention activity/assessment, 3) how well study participants complete each assessment (adherence to the intervention), and 4) what proportion of enrolled patients complete the intervention. Through this pilot study, the investigators will assess if the proposed intervention is acceptable to Hispanic kidney and liver cancer patients.

Additionally, the investigators will evaluate the effect of social support intervention on timely treatment initiation after diagnosis. Timely treatment after diagnosis will be based on time in days between cancer diagnosis with CT or MRI to initiation of definitive treatment (e.g., surgery, liver transplant, or ablation). Many kidney and liver cancer patients initiate treatment within 3 months after the diagnosis and continue to have follow-up care. Kidney cancer patients undergo an imaging assessment for other reasons and have incidental findings of a kidney mass. Adherence to follow-up care will be assessed based on whether patients schedule and show up for follow-up imaging assessment or scheduled appointments with hepatologists or urologists and how long the delay in the follow-up care is.

Intervention materials will be adapted from an existing, manualized symptom management intervention shown to be effective in reducing symptom burden in cancer survivors. Drs. Batai and Valencia will supervise the revision, translation, cultural adaptation, and illustration of the intervention to be linguistically and culturally appropriate for Spanish-speaking cancer survivors and caregivers. Intervention education materials will serve as an evidence-based guide for easy reference, including frequently asked questions, information on when to contact the health care provider (when patients have symptoms), strategies for communication with health care providers, family members and friends, and information on lifestyle modification (i.e. diet and physical activity) for cancer patients.

The results of this pilot intervention will be used to develop a larger, adequately-powered randomized controlled trial to robustly evaluate the effects of integrating existing social networks into care to reduce the negative effect of social deprivation and improve timeliness of treatment initiation and adherence to recommended treatment.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be adult Hispanic patients (age 18 or older) who have diagnosis of primary kidney and liver cancer through imaging assessment with CT or MRI at BUMC.

For liver cancer, we will include only HCC patients.

Exclusion Criteria:

* Patients with a small kidney mass (clinical T1a) who are undergoing active surveillance and patients with metastatic kidney or liver cancer will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Screening and enrollment figures | Screening and enrollment
  Screening and enrollment figures will be assessed as the number of patients who are screened and enrolled per month, respectively.
Study retention | 6-months post enrollment (end of the intervention)
  Retention will be assessed as the number of patients who complete the 6-month intervention activities and assessment in both the usual care control and intervention group.
Completeness of data collection | 9-months post enrollment
  Completeness of data collection will be assessed as the proportion of randomized patients who complete each study assessment, including any follow-up assessments.
Participant adherence to the intervention | 6-months post enrollment (end of intervention)
  The proportion of patients randomized to the intervention group who complete each of the 7 telephone sessions.
Acceptability of the intervention | 9-months post enrollment
  Patients' overall experience and satisfaction with the intervention, navigator's assessment of the overall impact of the intervention on secondary outcomes.

SECONDARY OUTCOMES:
Mean and median time to treatment initiation in the control vs. intervention group | 6-months post enrollment (end of intervention) and 12-months
  Time in days between the date of the liver or kidney cancer diagnosis (the date a CT or MRI was conducted that led to an abnormal finding) and the date of initiation of surgical treatment, liver transplant or ablation (whichever came first) in intervention compared to control group
Proportion of patients who attend a follow-up imaging assessment after their surgery with hepatologists or urologists in control vs. intervention group | 6-months post enrollment (end of intervention), 12-months, and 18-months
  Proportion of patients who receive the recommended post-surgical imaging (CT/MRI) assessment in intervention compared to control group
Proportion of patients who attend a scheduled appointment after their surgery with hepatologists or urologists in control vs. intervention group | 6-months post enrollment (end of intervention), 12-months, and 18-months
  Proportion of patients who attend a post-operative follow-up appointment in intervention compared to control group

CONTACTS AND LOCATIONS:
Overall Officials: Ken Batai, PhD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No